CLINICAL TRIAL: NCT05908838
Title: Randomized Clinical Trial:Clinical Study of Modified Banxia Xiexin Decoction Treatment on Gastric Cancer
Brief Title: Clinical Study of Modified Banxia Xiexin Decoction Treatment on Gastric Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: ShuGuang Hospital (Other)
Responsible Party: Principal Investigator, Mingyu Sun, Clinical Professor, ShuGuang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 42507214-11
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Gastric Cancer (Diagnosis)
Keywords: Modified Banxia Xiexin Decoction; Gastric Cancer; Clinical Efficacy; Randomized clinical trial; Mechanism
MeSH Terms: conditions — Stomach Neoplasms; Disease | interventions — Drug Therapy, Combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combination chemotherapy with Modified Banxia Xiexin Decoction (Active Comparator): 146 patients with gastric cancer were randomly divided into a treatment group of 73 cases and a control group of 73 cases. The treatment group received combination chemotherapy with Modified Banxia Xiexin Decoction
  Interventions: Drug: Modified Banxia Xiexin Decoction
- combination chemotherapy with Placebo granules (Placebo Comparator): The control group received combination chemotherapy with Placebo granules.
  Interventions: Drug: combination chemotherapy with Placebo granules

INTERVENTIONS:
Drug: Modified Banxia Xiexin Decoction — The treatment group#Modified Banxia Xiexin Decoction group#was given Modified Banxia Xiexin Decoction, 2 bags each time, 2 times a day, and 1 hour after meals. The control group(chemotherapy group)#Chemotherapy regimen was based on the Chinese Clinical Oncology Association Guidelines for the Diagnosis and Treatment of Gastric Cancer (2018), including oxaliplatin +5-FU/CF, SOX regimen, XELOX regimen, and S-1 monotherapy regimen.
  Arms: combination chemotherapy with Modified Banxia Xiexin Decoction
Drug: combination chemotherapy with Placebo granules — combination chemotherapy with Placebo granules
  Arms: combination chemotherapy with Placebo granules

SUMMARY:
Research purpose To elucidate the effect mechanism and clinical effective of Modified Banxia Xiexin Decoction in the prevention and treatment of gastric cancer. From genes related to cell differentiation, proliferation, apoptosis, tumor invasion and metastasis, genes related to immune inflammation and immune escape and other possible aspects to elucidate the effective and mechanism of Modified Banxia Xiexin Decoction's treatment on gastric cancer

DETAILED DESCRIPTION:
Modified Banxia Xiexin Decoction treatment and mechanism on Gastric Cancer. Main Responsibility Person: Mingyu Sun research center#Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine Trial Objective#Observe the clinical efficacy and mechanism of Modified Banxia Xiexin Decoction in the treatment gastric cancer Therapeutic Schedule#In this study, 146patients with gastric cancer who received chemotherapy in the Department of Gastrointestinal Surgery and Oncology, Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine were recruited and divided into groups according to random number table method, namely, 73 patients in the Modified Banxia Xiexin Decoction combined chemotherapy group and 73 patients in the Placebo granules combined chemotherapy group.Modified Banxia Xiexin Decoction group was treated with 18 weeks of Chinese patent medicine Modified Banxia Xiexin Decoction at the same time of chemotherapy. The Overall survival, Progression-free survival, Solid tumor efficacy, TCM syndrome score, quality of life score, Tumor markers, Immune function and adverse reactions of the two groups before and 18 weeks after treatment were observed and compared. Elucidate the possible mechanism of action of Modified Banxia Xiexin Decoction in the treatment of gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage IV gastric cancer with a clear cytological or pathological diagnosis.
2. The patient is willing to receive palliative chemotherapy (more than 6 months between the first treatment or the last chemotherapy).
3. At least one measurable lesion revealed by imaging (PET-CT, CT, MRI, bone scan, x-ray).
4. Expected survival of ≥ 6 months.
5. It is consistent with the diagnosis of spleen qi deficiency and cold-heat mismatch in TCM.
6. Age 18 to 75 years with a physical condition score of ECOG (0-1).
7. The blood count is normal, heart, liver and kidney functions are not abnormal, and the electrocardiogram is basically normal.
8. Patients have good compliance, are able to understand the study and sign an informed consent form.

Exclusion Criteria:

1. Those with a history of severe cardiovascular, urinary, hematological and digestive system diseases.
2. Pregnant or breastfeeding women with uncontrollable mental disorders.
3. With gastrointestinal obstruction or active bleeding in the gastrointestinal tract, as well as perforation and dysphagia.
4. Complications of serious infectious diseases such as active tuberculosis.
5. Those with contraindications to chemotherapy or frequent vomiting.
6. Poor compliance.
7. Patients who have used other trial drugs or in other clinical trials in the past month.

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Overall survival | the patients' were included into the clinical trials and up to 18 weeks treatment
  To observe the effects of treatment group and control group on OS in patients with advanced gastric cancer, and evaluate whether there is statistical difference in OS between the two groups.From date of randomization until the date of death from any cause, whichever came first, assessed up to 18 months.

SECONDARY OUTCOMES:
Progression-free survival | the patients' were included into the clinical trials and up to 18 weeks treatment
  The time between the first treatment and tumor progression or death.From date of randomization until the date of first documented progression, whichever came first, assessed up to 18 months. To observe the effects of treatment group and control group on PFS in patients with advanced gastric cancer, and evaluate whether there is a statistical difference in PFS between the two groups.
EORTC QLQ-C30 | the patients' were included into the clinical trials and up to 18 weeks treatment
  The quality of life score is based on the EuroPean organization for Research and Treatment (EORTC) Quality of Life Scale (QLQ-C30 v3.0), which records changes in quality of life before and after treatment and compares them. Linear transformation of statistical results was performed to obtain standardized scores (0~100 points), so that scores in various fields could be compared with each other, and the problem of reverse entries could be solved at the same time. The higher the score of symptom field obtained by each subscale, the worse the quality of life condition. The higher the scores in the areas of function and general health, the better the patient's quality of life. Analyze whether there was a statistical difference between the two groups.
Clinical symptoms | the patients' were included into the clinical trials and up to 18 weeks treatment
  According to the scoring criteria of the Guidelines for Clinical Research of New Chinese Medicines (2002), the symptoms of patients after treatment were determined. The improvement of patients' overall symptoms was evaluated by Nimodipine method, and the efficacy index after treatment = (total score before treatment - total score after treatment)/total score before treatment *100%.
Tumor markers | the patients' were included into the clinical trials and up to 18 weeks treatment
  Detect the biomarkers (CA72-4, CEA, CA19-9, CA242, CA50, CA125) of two groups of patients before and after treatment to determine whether there is a statistical difference between the two groups before and after treatment.
Immune function | the patients' were included into the clinical trials and up to 18 weeks treatment
  T cell subsets of the two groups to determine whether there was a statistical difference between the two groups before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mingyu Sun, doctor, Principal Investigator — Ethics Committee of Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: Undecided